CLINICAL TRIAL: NCT00815126
Title: Association Between Nasal Provocation Test With Lysine-Acetylsalicylate(ASA) and Clinical Diagnosis in Patients With Aspirin/Nonsteroidal Anti-Inflammatory Drugs(NSAIDs) and/or Acetaminophen Immediate Sensitivity Reactions
Brief Title: Nasal Provocation Test With Lysine-Acetylsalicylate (ASA) in Patients With Nonsteroidal Anti-Inflammatory Drugs (NSAIDs) Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Jettanong Klaewsongkram, MD, Chulalongkorn University
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Chula-ARC 002/08
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Aspirin Hypersensitivity; NSAIDs Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mucocutaneous symptoms from NSAIDs (Active Comparator)
  Interventions: Procedure: Lysine-ASA Nasal ProvocationTest
- Respiratory symptoms from NSAIDs (Active Comparator)
  Interventions: Procedure: Lysine-ASA Nasal ProvocationTest
- NSAIDs tolerant individuals (Active Comparator)
  Interventions: Procedure: Lysine-ASA Nasal ProvocationTest

INTERVENTIONS:
Procedure: Lysine-ASA Nasal ProvocationTest — Lysine-ASA 80 µl (16 mg of aspirin) will be installed in both nostrils with pipette

SUMMARY:
This study aims to compare the efficacy of nasal provocation test with Lysine-Acetylsalicylate in patients with history of NSAIDs hypersensitivity between mucocutaneous symptoms and respiratory symptoms and laboratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of ASA/NSAIDs hypersensitivity with mucocutaneous symptoms and/or respiratory symptoms

Exclusion Criteria:

* Patients who cannot discontinue drugs before the test as follow

  * Nasal corticosteroids/Oral corticosteroids/Leukotriene modifiers for 1 week
  * Short-acting antihistamines for 3 days
  * Nasal a-mimetics/Oral a-mimetics/Local cromones for 24 hours
* Contraindicated for nasal provocation test: pregnant, exacerbation of allergic rhinitis/asthma, having upper respiratory tract infection within 2 weeks prior to the test, having nose surgery within 8 weeks prior to the test, having severe systemic disease(s)
* Having factors interfere nasal provocation test with Lysine-ASA such as massive nasal polyp, nasal septal perforation, total nasal obstruction at least 1 nostril

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Symptom scores and/or acoustic rhinometry result upon Lysine-ASA nasal provocation test in patients with history of mucocutaneous or respiratory symptoms from NSAIDs | 5 months

SECONDARY OUTCOMES:
Correlation between clinical manifestations and laboratory results (basophil activation test, etc.) | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand